CLINICAL TRIAL: NCT02136446
Title: Prospective Post-market Evaluation of an Echogenic Catheter Used in a Peripheral Nerve Block Procedure
Brief Title: Prospective Post-market Evaluation of an Echogenic Catheter
Acronym: EchoCath
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Smiths Medical, ASD, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EchoCath
Record Dates: First submitted 2014-05-07; First posted 2014-05-13 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Peripheral Nerve Block Procedure
Keywords: Paravertebral block; Mastectomy; Post-operative pain; Echogenic; Peripheral nerve block catheter
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EchoGlo™ Peripheral Nerve Block Catheter (Experimental): Echogenic nerve block catheter (test)
  Interventions: Device: EchoGlo Nerve Block Catheter
- Pajunk® EpiLong Catheter (Active Comparator): Non-echogenic nerve block catheter (control)
  Interventions: Device: Pajunk® Nerve Block Catheter

INTERVENTIONS:
Device: EchoGlo Nerve Block Catheter — Catheter used for a paravertebral anesthesia block
  Other Names: EchoGlo™ Peripheral Nerve Block Catheter
  Arms: EchoGlo™ Peripheral Nerve Block Catheter
Device: Pajunk® Nerve Block Catheter — Nerve Block Catheter
  Other Names: Pajunk® EpiLong Catheter
  Arms: Pajunk® EpiLong Catheter

SUMMARY:
Patients scheduled for mastectomy and suitable for paravertebral block will be randomized to one of 2 groups.

Group 1 will have the nerve block performed using a standard non-echogenic needle and catheter under ultrasound guidance. Group 2 will have the block performed using the control needle and an echogenic catheter, all under ultrasound (US) guidance.

The clinician will be blinded to the catheter type and will assess the quality of catheter visualisation of the US image during the procedure, along with adequacy of spread of local anesthetic. The primary outcome will be needle visibility, and secondary outcomes will be block success rate and block quality. An assessment of the patient's pain levels after the procedure will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo breast surgery requiring use of a peripheral nerve block catheter for establishing a paravertebral block
* Patients classified as ASA (American Society of Anesthesiologists) physical status I, II or III
* Patients at least 18 years old
* Patient is willing and able to provide informed consent for study participation
* Patient has a good understanding of written and verbal English

Exclusion Criteria:

* Patient with contraindications to regional anesthesia technique (e.g. allergy to local anesthetic or other medications used in study)
* Patient with known coagulopathy
* Patient whose target nerve cannot be seen with linear ultrasound probe in a pre-procedure scan. All patients who need a curvilinear probe to visualize the target nerve will be excluded from the study.
* Patients having mastectomy and immediate reconstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Visibility of entire catheter length | Day 1, time of procedure
  Demonstrate superior ultrasound visibility of the entire length of the test catheter compared to the control, as graded by a blinded investigator
Visibility of catheter tip | Day 1, time of procedure
  Demonstrate superior ultrasound visibility of the test catheter tip compared to the control, as graded by a blinded investigator

SECONDARY OUTCOMES:
Quality of the block | Day 1, time of procedure
  Mean rating of block quality as assessed by the clinician on a 4 point scale per treatment group
Block failure rate | Day 1, time of procedure
  Number of failed blocks per treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Kratz, MS, Study Director — Smiths Medical
Locations (1):
- University College Hospital, London, United Kingdom